CLINICAL TRIAL: NCT00507936
Title: A Global, Multicenter, Randomized, Double-Blind Placebo Controlled Study Comparing the Safety and Efficacy of ABT-894, Duloxetine and Placebo in Subjects With Diabetic Neuropathic Pain
Brief Title: Safety and Efficacy Study in Subjects With Diabetic Neuropathic Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M06-850; 2007-001139-71 (EudraCT Number)
Record Dates: First submitted 2007-07-25; First posted 2007-07-27 (Estimated); Last update posted 2013-01-23 (Estimated); Status verified 2013-01

CONDITIONS: Diabetic Neuralgia; Diabetic Neuropathies; Diabetic Neuropathy, Painful; Diabetic Polyneuropathy; Neuralgia, Diabetic
Keywords: Diabetic Neuropathy; Painful; Diabetic Polyneuropathy; Neuralgia; Diabetic; Diabetic Neuropathies; Diabetic Neuralgia
MeSH Terms: conditions — Diabetic Neuropathies; Pain; Neuralgia | interventions — 3-(5,6-dichloropyridin-3-yl)-3,6-diazabicyclo(3.2.0)heptane; Duloxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- A (Experimental): ABT-894 1 mg BID
  Interventions: Drug: ABT-894
- B (Experimental): ABT-894 2 mg BID
  Interventions: Drug: ABT-894
- C (Experimental): ABT-894 4 mg BID
  Interventions: Drug: ABT-894
- D (Placebo Comparator)
  Interventions: Drug: placebo
- E (Active Comparator): Duloxetine 60 mg QD
  Interventions: Drug: Duloxetine

INTERVENTIONS:
Drug: ABT-894 — ABT-894 1 mg capsule BID throughout treatment period
  Arms: A
Drug: ABT-894 — ABT-894 2 mg capsule BID throughout treatment period
  Arms: B
Drug: ABT-894 — ABT-894 4 mg capsule BID throughout treatment period
  Arms: C
Drug: placebo — placebo capsule BID throughout the treatment period
  Arms: D
Drug: Duloxetine — Duloxetine 60 mg QD throughout treatment period
  Arms: E

SUMMARY:
This study will compare the efficacy and the safety of ABT-894 (1mg, 2mg or 4mg capsules) administered BID to placebo in the treatment of DNP. Another treatment arm will be Duloxetine 60mg administered once daily (QD). Approximately 275 subjects will be enrolled into the study at approximately 50 sites in both the United States and Europe. The study will be divided into the following periods: Screening/Washout (21 days) followed by a Baseline Visit, an 8-week Treatment Period and a 1-week Follow-up Visit.

ELIGIBILITY:
Inclusion Criteria:

* If female, subject is either postmenopausal for at least two (2) years or surgically sterile or is practicing at least one (1) method of birth control.
* If female, subject must have negative results for pregnancy tests.
* The subject must have a diagnosis of diabetes mellitus (Type 1 or Type 2) and a diagnosis of DNP.
* Subject's DNP must be present for a minimum of six (6) months and should have begun in the feet with relative symmetrical onset.
* Subject has an HgbA1c <= 9. Subjects who have an HgbA1c > 9 and <= 11 may be included in the study.
* If male, the subject is surgically sterile (vasectomy), is sexually inactive, or is using a barrier method (condom) of birth control for the duration of the study and for 7 days following the last dose of study drug.

Exclusion Criteria:

* The subject has failed previous treatment with duloxetine for DNP.
* Subject has a diagnosis of narrow-angle glaucoma.
* Subject has a history of an allergic reaction or intolerance to duloxetine, acetaminophen, or any other NNR agonist.
* Subject has a diagnosis of fibromyalgia that requires treatment.
* Subject has a functioning implanted medical device (spinal cord stimulator, intrathecal pump or peripheral nerve stimulator) for the treatment of neuropathic pain.
* Subject has a history of seizures (febrile may be ok) or major depressive episode within the past two (2) years or major psychiatric disorder including bipolar disorder, schizophrenia or borderline personality disorder.
* Subject has a history of myocardial infarction (MI) within six (6) months of the Screening Visit.
* Subject has unstable angina.
* Subject has ventricular arrhythmia requiring anti-arrhythmic therapy.
* Subject has undergone a cardiac revascularization procedure within 30 days of Screening.
* Subject has uncontrolled hypertension (HTN) defined as a systolic blood pressure (BP) >= 160 and/or a diastolic blood pressure (BP) >= 100 at Screening and/or Baseline.
* Subject has a clinically significant abnormal ECG at Screening
* Subject has an active malignancy of any type or has been diagnosed with or treated for cancer within the past 5 years.
* Subject has a positive result for drugs of abuse at Screening with the exception of a positive result for a known prescribed medication.
* Subject's screening laboratory results show hepatitis A, B or C.
* Subject has a known or suspected history of Human Immunodeficiency Virus (HIV).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2007-08; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Efficacy of each ABT-894 dose (1 mg, 2 mg, or 4 mg BID) versus placebo in the treatment of pain due to DNP | Change from baseline to final 24-hour average pain score

SECONDARY OUTCOMES:
Proportions of treatment responders; subjects who complete treatment period with 30% improvement | From Baseline to final 24-hour average pain score
Mean of 24-hour worst pain severity, average of night pain, and average of morning pain measured by the 11-point Likert scale and from subject's daily diary | Weekly through treatment phase
Brief Pain Inventory (BPI) (short form) including Pain Severity | At each visit from Baseline to Week 8 visit
Clinician Global Impression: Severity (CGI-S) and Patient Global Impression: Change (PGI-C) | At each visit from Baseline to Week 8 visit

CONTACTS AND LOCATIONS:
Overall Officials: Wolfram Nothaft, MD, Study Director — AbbVie
Locations (49):
- United States (29):
  - Site Reference ID/Investigator# 5207, Mesa, Arizona
  - Site Reference ID/Investigator# 6053, Phoenix, Arizona
  - Site Reference ID/Investigator# 5206, Little Rock, Arkansas
  - Site Reference ID/Investigator# 7387, North Little Rock, Arkansas
  - Site Reference ID/Investigator# 6052, Anaheim, California
  - Site Reference ID/Investigator# 7064, Garden Grove, California
  - Site Reference ID/Investigator# 8286, National City, California
  - Site Reference ID/Investigator# 5276, Clearwater, Florida
  - Site Reference ID/Investigator# 6781, Hialeah, Florida
  - Site Reference ID/Investigator# 7514, Palm Beach Gardens, Florida
  - Site Reference ID/Investigator# 8113, Tampa, Florida
  - Site Reference ID/Investigator# 6047, Pasadena, Maryland
  - Site Reference ID/Investigator# 5277, Brockton, Massachusetts
  - Site Reference ID/Investigator# 6043, St Louis, Missouri
  - Site Reference ID/Investigator# 6044, St Louis, Missouri
  - Site Reference ID/Investigator# 7906, Omaha, Nebraska
  - Site Reference ID/Investigator# 6045, New York, New York
  - Site Reference ID/Investigator# 5946, New York, New York
  - Site Reference ID/Investigator# 5216, New York, New York
  - Site Reference ID/Investigator# 7483, New York, New York
  - Site Reference ID/Investigator# 5947, Cincinnati, Ohio
  - Site Reference ID/Investigator# 6869, Cuyahoga Falls, Ohio
  - Site Reference ID/Investigator# 5217, Portland, Oregon
  - Site Reference ID/Investigator# 7699, Houston, Texas
  - Site Reference ID/Investigator# 5836, San Antonio, Texas
  - Site Reference ID/Investigator# 5899, San Antonio, Texas
  - Site Reference ID/Investigator# 5950, San Antonio, Texas
  - Site Reference ID/Investigator# 7187, San Antonio, Texas
  - Site Reference ID/Investigator# 6054, Seattle, Washington
- Canada (3):
  - Site Reference ID/Investigator# 8508, Kingston
  - Site Reference ID/Investigator# 8436, Laval
  - Site Reference ID/Investigator# 8481, Winnipeg
- France (5):
  - Site Reference ID/Investigator# 5258, Corbeil-Essonnes
  - Site Reference ID/Investigator# 7696, Nanterre
  - Site Reference ID/Investigator# 5260, Narbonne
  - Site Reference ID/Investigator# 5171, Nevers
  - Site Reference ID/Investigator# 7115, Nîmes
- Germany (5):
  - Site Reference ID/Investigator# 6763, Berlin
  - Site Reference ID/Investigator# 7117, Essen
  - Site Reference ID/Investigator# 5034, Frankfurt
  - Site Reference ID/Investigator# 6760, Heidelberg
  - Site Reference ID/Investigator# 6732, Mainz
- Italy (2):
  - Site Reference ID/Investigator# 5018, Milan
  - Site Reference ID/Investigator# 5006, Rome
- Mexico (3):
  - Site Reference ID/Investigator# 8427, Guadalajara
  - Site Reference ID/Investigator# 8497, Mexico City
  - Site Reference ID/Investigator# 8125, Monterrey, N.L.
- Puerto Rico (2):
  - Site Reference ID/Investigator# 8120, Ponce
  - Site Reference ID/Investigator# 8121, San Juan